CLINICAL TRIAL: NCT02960295
Title: The Virtual Visit for Women With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10539
Record Dates: First submitted 2016-10-18; First posted 2016-11-09 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual visit (Experimental): 1. Self-monitoring of blood glucose (four times daily).
  2. Self-weighing (weekly).
  3. Self-checking of blood pressure (weekly).
  4. Checking fetal heart rate (weekly).
  5. Visits with caregivers.
  Interventions: Device: 1-Self-monitoring of blood glucose; Device: 2-Self-weighing; Device: 3-Self-checking of blood pressure; Device: 4-Checking fetal heart rate; Procedure: 5-Visits with caregivers

INTERVENTIONS:
Device: 1-Self-monitoring of blood glucose — Self-monitoring of blood glucose 4 times daily: fasting and 1-hour after each meal. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment. Intervention: At every office visit and at every telephone ("virtual") visit the patient's physician will review glucose results and make adjustments in diet, activity, or medication to bring glucose into desired range.
Device: 2-Self-weighing — Self-weighing on electronic scale at least once a week. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment. Consultation with the nutritionist will be obtained for women gaining in excess of or less than that indicated for her pre-pregnancy BMI, per Institute of Medicine (IOM) standards.
Device: 3-Self-checking of blood pressure — Self-checking of blood pressure at least weekly with sphygmomanometer. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment. Patients with elevated blood pressure will be requested to come to Obstetrics Triage immediately for further assessment.
Device: 4-Checking fetal heart rate — Patient will record her fetus' heart rate with a Doppler device at least once weekly. The patient will immediately report to Labor and Delivery for any fetal heart rate below 100 beats per minute or greater than 160 beats per minute over a 10 minute observation period.Those reporting a fetal heart rate outside of the normal range will be requested to come to ObstetricTriage for further assessment.
Procedure: 5-Visits with caregivers — Telephone visits will alternate with in-office visits.Those failing to keep appointments will be contacted and reappointed at a mutually convenient time.

SUMMARY:
This is a feasibility study of care for women with gestational diabetes (GDM) using electronic equipment to participate in virtual office visits.

Participants will be trained in the use of glucose meters, scales, and sphygmomanometers which are Bluetooth connected to an app on their cellphones. Fetal well-being will be assessed with Dopplers and kick counts. Care will be delivered by alternate in-office and telephone visits.

DETAILED DESCRIPTION:
The core elements of a prenatal visit for any pregnant woman include assessment of BP, weight, and presence of fetal heart activity. The treatment of GDM additionally requires the measurement of and review of maternal glycemia. Technology exists for patients to measure these parameters and to relay this information securely directly from these devices via the internet to the healthcare provider's office. A key element of antepartum care for GDM, self-monitoring of blood glucose (SMBG), has for some years been conducted with memory-based portable glucose meters. To assure accuracy in reports of patient measurements, it is important that all devices be of a design wherein results of measures of patient parameters are transmitted in unedited fashion directly devices to the health care provider. While no data exists about the accuracy of self-reporting of patient weight and blood pressure, intentional or unintentional alteration in reports of self-monitored glucose results is a known risk of reliance on patient self-reported data. This pilot study will explore the feasibility of the use of this technology from patients' homes in lieu of an office visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of gestational diabetes
2. Singleton pregnancy
3. <32 weeks gestation
4. Age 18-45 years
5. Fluent and literate in English or Spanish
6. Have a cellphone with capability of internet access.

Exclusion Criteria:

1. Multiple gestations (twins or higher)
2. Have a history of fetal demise
3. Have a history of chronic health problems that might affect outcomes (such as HIV, treatment with steroids, significant cardiac or renal disease, or chronic hypertension), and those who had bariatric surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women meeting inclusion and exclusion criteria (see below) who volunteer to participate for the study. Volunteers will be solicited sequentially.
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Sacks, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Given JE, Bunting BP, O'Kane MJ, Dunne F, Coates VE. Tele-Mum: A Feasibility Study for a Randomized Controlled Trial Exploring the Potential for Telemedicine in the Diabetes Care of Those with Gestational Diabetes. Diabetes Technol Ther. 2015 Dec;17(12):880-8. doi: 10.1089/dia.2015.0147. Epub 2015 Sep 22. PMID 26394017
- [Result] Homko CJ, Deeb LC, Rohrbacher K, Mulla W, Mastrogiannis D, Gaughan J, Santamore WP, Bove AA. Impact of a telemedicine system with automated reminders on outcomes in women with gestational diabetes mellitus. Diabetes Technol Ther. 2012 Jul;14(7):624-9. doi: 10.1089/dia.2012.0010. Epub 2012 Apr 18. PMID 22512287
- [Derived] Sacks DA, Ling Grant D, Macias M, Li X, Lawrence JM. The Virtual Office Visit for Women With Gestational Diabetes Mellitus. Diabetes Care. 2017 Mar;40(3):e34-e35. doi: 10.2337/dc16-2569. Epub 2017 Jan 11. No abstract available. PMID 28077459

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Visit: Pregnant women with gestational diabetes (GDM) who will:
  1-self-monitor blood glucose 4 times daily, 2-self-weigh themselves weekly, 3-self-check their blood pressure weekly, 4-check their fetus' heart rate weekly, and 5-alternate office visits with telephone visits with their caregivers
  1. Self-monitoring of blood glucose: Self-monitoring of blood glucose 4 times daily: fasting and 1-hour after each meal. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  2. Self-weighing: Self-weighing on electronic scale at least once a week. Results will be transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  3. Self-checking of blood pressure: Self-checking of blood pressure at least weekly with sphygmomanometer. Results will be transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  4. Checking fetal
Period: Overall Study
Arm/Group | Virtual Visit
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pregnant women with gestational diabetes
Groups:
- Virtual Visit: Pregnant women with GDM who will:
  1-self-monitor blood glucose four times daily, 2-self-weigh themselves weekly, 3-self-check their blood pressure weekly, 4-check their fetus' heart rate weekly, and 5-alternate office visits with telephone visits with their caregivers
  1. Self-monitoring of blood glucose: Self-monitoring of blood glucose 4 times daily: Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  2. Self-weighing: Self-weighing on electronic scale at least once a week. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  3. Self-checking of blood pressure: Self-checking of blood pressure at least weekly with sphygmomanometer. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  4. Checking fetal
Arm/Group | Virtual Visit
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, in years, was collected upon enrollment for the study
  years | 30 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were pregnant women
  Participants
    Female | 10
    Male | 0
Compliance with requirements of study [Count of Participants; unit: Participants] — Number of participants who met all the eligibility criteria required to participate in the study
  Participants | 10

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Requirements for Frequency of Glucose Measures
Description: Each patient is requested to check her blood glucose four times a day: fasting and one hour after the first bite of each meal. Compliance with this requirement will be measured for each patient by dividing the number of daily glucose checks actually performed by the number of days in the study.
Time Frame: 1 year
Population: women with gestational diabetes
Measure: Mean (Standard Deviation); unit: number of glucose checks per pt per day
Groups:
- Virtual Visit: all participants
Arm/Group | Virtual Visit
Number analyzed (Participants) | 10
number of glucose checks per pt per day | 3.1 (1.26)
Statistical Analysis 1: Comparison: Virtual Visit; In this interventional study the number of glucose checks per patient per day was calculated as stated above. There was no comparison group and no test of statistical significance; Test type: Other — There was no comparison group and no test of statistical significance; This is a simple calculation of the mean (sd) of the number of glucose checks per pt per day

2. Secondary Outcome: Compliance With Self-weighing Requirements
Description: Average percentage of weight checks per week in study, calculated as total weight checks in study/weeks in study x 100
Time Frame: 1 year
Population: Women with gestational diabetes
Measure: Mean (Standard Deviation); unit: percentage of weekly weights performed
Groups:
- Virtual Visit: 1-Self-monitoring of blood glucose (four times daily). 2-Self-weighing (weekly). 3-Self-checking of blood pressure (weekly). 4-Checking fetal heart rate (weekly). 5-Visits with caregivers.
  1. Self-monitoring of blood glucose: Self-monitoring of blood glucose 4 times daily: fasting and 1-hour after each meal. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment. Intervention: At every office visit and at every telephone ("virtual") visit the patient's physician will review glucose results and make adjustments in diet, activity, or medication to bring glucose into desired range.
  2. Self-weighing: Self-weighing on electronic scale at least once a week. Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment. Consultation with the nutritionist will be obtained for women gaining in excess of or less than that indicated for her
Arm/Group | Virtual Visit
Number analyzed (Participants) | 10
percentage of weekly weights performed | 136 (76)
Statistical Analysis 1: Comparison: Virtual Visit; Test type: Other — This is an observational study; p < 0.05, Pearson correlation (r)
Statistical Analysis 2: Comparison: Virtual Visit; Test type: Other — This is an observational study; p < 0.05, Pearson correlation coefficient (r)
Statistical Analysis 3: Comparison: Virtual Visit; Test type: Other; p < 0.05, Pearson correlation coefficient (r)

3. Secondary Outcome: Compliance With Blood Pressure Checking Requirements
Description: Percentage of required once-weekly blood pressure checks calculated as total blood pressure checks in study/weeks in study x 100
Time Frame: 1 year
Population: Percentage of required once-weekly blood pressure checks calculated as total blood pressure checks in study/weeks in study x 100
Measure: Mean (Standard Deviation); unit: percentage of Blood Pressure checks
Arm/Group | Virtual Visit
Number analyzed (Participants) | 10
percentage of Blood Pressure checks | 162.5 (69.48)

4. Secondary Outcome: Glucose Concentrations
Description: Mean of all glucose measures during study, in mg/dl
Time Frame: 1 year
Population: Mean of all glucose measures during study, in mg/dl
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Virtual Visit
Number analyzed (Participants) | 10
milligrams per deciliter | 106.0 (3.83)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Definitions used were those of clinicaltrials.gov.
Groups:
- Virtual Visit: Pregnant women with GDM who will:
  1-self-monitor blood glucose four times daily, 2-self-weigh themselves weekly, 3-self-check their blood pressure weekly, 4-check their fetus' heart rate weekly, and 5-alternate office visits with telephone visits with their caregivers
  1. Self-monitoring of blood glucose: Self-monitoring of blood glucose 4 times daily: Results will be recorded and transmitted in real-time via a Bluetooth connection to a cellphone app installed on study enrollment.
  2. Self-weighing: Self-weighing on electronic scale at least once a week.
  3. Self-checking of blood pressure: Self-checking of blood pressure at least weekly with sphygmomanometer.
  4. Checking fetal heart rate: Patient will record her fetus' heart rate with a Doppler device at least once weekly.
  5. Visits with caregivers: Telephone visits will alternate with in-office visits
Arm/Group | Virtual Visit
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes